CLINICAL TRIAL: NCT01109355
Title: Effect of Positive End Expiratory Pressure on Cerebral Perfusion Pressure in Adult Patients With Hemorrhagic Stroke
Brief Title: Positive and Expiratory Pressure and Hemorrhagic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Wildberg Alencar, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Berg 01
Record Dates: First submitted 2010-04-19; First posted 2010-04-23 (Estimated); Last update posted 2010-04-23 (Estimated); Status verified 2009-12

CONDITIONS: Stroke; Hemorrhage
Keywords: PEEP; Patients with hemorrhage stroke under mechanical ventilation
MeSH Terms: conditions — Stroke; Hemorrhage | interventions — Hemodynamics; Intracranial Pressure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: lung mechanics ventilatory — To perform the evaluation of lung mechanics ventilatory mode was changed to control volume with the following parameters: tidal volume (Vt) = 8ml/kg weight, peak flow (PF) = 6 x minute volume, fraction of inspired O2 (FiO2) = 40%, respiratory rate (RR) = 16 bpm, sensitivity = 1 cmH2O. The following variables were monitored: PIC, Blood Pressure (BP), heart rate (HR), peak pressure in the airways (pp.) and plateau pressure of the respiratory system (Ppl.), these values were monitored with PEEP = 5 cmH2O. PEEP employed ranged from 0 to 14 cmH2O. To eliminate a possible physiological accommodation by the progressive increase of PEEP, the range of values was determined by drawing a sealed envelope for each patient, ranging from 2 to 2 cmH2O.
Other: Hemodynamic and intracranial pressure — At each value of PEEP the patient was ventilated for a period of five minutes to carry out monitoring of ICP, BP, HR, PPC and peripheral oxygen saturation (SpO2). The ICP monitoring catheter was kept closed for drainage and open for monitoring, since the arrival of the surgical block, was only open for drainage if there was an increase in ICP above 20 mmHg.

SUMMARY:
Intrathoracic positive pressure may lead to a change hemodynamics, with repercussions for the intracranial compartment, thereby altering intracranial pressure (ICP) and cerebral perfusion pressure (CPP). This effect may become more intense when using high positive end expiratory pressure (PEEP) values. The aim of the present study was to measure the impact of different PEEP values on ICP, CPP and mean arterial pressure (MAP). MAP, whereas high PEEP values increase ICP, although without clinical relevance.

DETAILED DESCRIPTION:
This study is a prospective clinical trial, developed in the neurological intensive care unit approved by the ethics committee and research in humans. The charge of each patient had information about the study through the completion of informed consent and signed him when he agreed. Were the following inclusion criteria: adult patients with acute CVA and presence of ventricular drainage catheter for invasive monitoring of ICP and without intracranial hypertension. Were adopted as exclusion criteria: increased intracranial pressure, hemodynamic instability as a criterion of loss was used to expressions of interest in charge to leave. All patients completed the study. <br>All patients were from the surgical implantation of the ventricular catheter, arriving to the ICU intubated orally and manually ventilated with an Ambu bag. Were subjected to routine procedures: adjusting the mechanical ventilator (Inter5, Intermed, BR) during assisted controlled cycled pressure and facility to monitor vital signs. After thirty minutes of stable ICU patient in a supine position with head elevated 30 °, the protocol was initiated to assess the impact of PEEP on ICP. To perform the evaluation of lung mechanics ventilatory mode was changed to control volume with the following parameters: tidal volume (Vt) = 8ml/kg weight, peak flow (PF) = 6 x minute volume, fraction of inspired O2 (FiO2) = 40%, respiratory rate (RR) = 16 bpm, sensitivity = 1 cmH2O. The following variables were monitored: PIC, Blood Pressure (BP), heart rate (HR), peak pressure in the airways (pp.) and plateau pressure of the respiratory system (Ppl.), these values were monitored with PEEP = 5 cmH2O. <br>During the assessment protocol was changed to pressure control ventilation mode with the following values of ventilatory parameters: Pp = 30 cm H2O, inspiratory time = 1s; FiO2 = 40%, RR = 16 bpm; Sensitivity = 1 cmH2O. PEEP employed ranged from 0 to 14 cmH2O. To eliminate a possible physiological accommodation by the progressive increase of PEEP, the range of values was determined by drawing a sealed envelope for each patient, ranging from 2 to 2 cmH2O. At each value of PEEP the patient was ventilated for a period of five minutes to carry out monitoring of ICP, BP, HR, PPC and peripheral oxygen saturation (SpO2). The ICP monitoring catheter was kept closed for drainage and open for monitoring, since the arrival of the surgical block, was only open for drainage if there was an increase in ICP above 20 mmHg. <br>The monitoring was carried out using the multiparameter monitor (Siemens 7000). For ICP monitoring the ventricular catheter was connected to a pressure transducer and this monitor. <br>After the parameters evaluated with seven different PEEP values, the ventilatory mode was changed again to control volume again to evaluate pulmonary mechanics with the same initial parameters.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with acute CVA
* presence of ventricular drainage catheter for invasive monitoring of ICP
* without intracranial hypertension.

Exclusion Criteria:

* intracranial hypertension
* hemodynamic instability.

Ages: 42 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-01; Primary Completion 2008-07 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Measurement of intracranial pressure
  The ICP monitoring catheter was kept closed for drainage and open for monitoring, since the arrival of the surgical block, was only open for drainage if there was an increase in ICP above 20 mmHg.

SECONDARY OUTCOMES:
Effect of different values of PEEP on lung mechanics
  - Lung compliance:During the assessment protocol was changed to pressure control ventilation mode with the following values of ventilatory parameters: Pp = 30 cm H2O, inspiratory time = 1s; FiO2 = 40%, RR = 16 bpm; Sensitivity = 1 cmH2O. PEEP employed ranged from 0 to 14 cmH2O.
Effect of different PEEP levels on aspects hemodynamic
  At each value of PEEP the patient was ventilated for a period of five minutes to carry out monitoring of heart rate and cerebral perfusion pressure(CPP).

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Campelo, Study Chair — Universidade Federal de Pernambuco
Locations (1):
- Hospital Português, Recife, Pernambuco, Brazil

REFERENCES:
- [Result] Pillai S, Praharaj SS, Rao GS, Kolluri VR. Cerebral perfusion pressure management of severe diffuse head injury: effect on brain compliance and intracranial pressure. Neurol India. 2004 Mar;52(1):67-71. PMID 15069242
- [Result] Mayer SA, Copeland D, Bernardini GL, Boden-Albala B, Lennihan L, Kossoff S, Sacco RL. Cost and outcome of mechanical ventilation for life-threatening stroke. Stroke. 2000 Oct;31(10):2346-53. doi: 10.1161/01.str.31.10.2346. PMID 11022062